CLINICAL TRIAL: NCT03405441
Title: A 2-Part, Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-55375515 in Healthy Male Subjects
Brief Title: A Study to Investigate Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-55375515 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR108409; 55375515EDI1002 (Other: Janssen Research & Development, LLC); 2017-002457-11 (EudraCT Number)
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Panel 1): JNJ-55375515 and placebo (Experimental): Participants will receive dose level (DL) 1 of JNJ-55375515 (starting dose) or placebo on Day 1 of period 1 based on their randomization sequence 1, 2 or 3. Dose of the study medication will be escalated to DL 3 (period 2) and a maximum of DL 5 (period 3) based on the safety and tolerability profile and pharmacodynamic (PD) profile assessed at the preceding dose level. A wash-out period of at least 10 days will be maintained between study drug administrations.
  Interventions: Drug: JNJ-55375515 Dose Level 1; Drug: JNJ-55375515 Dose Level 3; Drug: JNJ-55375515 Dose Level 5; Drug: Placebo
- Part 1 (Panel 2): JNJ-55375515 and placebo (Experimental): Participants will receive DL 2 of JNJ-55375515 (starting dose) or placebo on Day 1 of period 1 based on their randomization sequence 1, 2 or 3. Dose of the study medication will be escalated to DL 4 (period 2) and a maximum of DL 6 (period 3) based on the safety and tolerability profile and PD profile assessed at the preceding dose level. A wash-out period of at least 10 days will be maintained between study drug administrations.
  Interventions: Drug: JNJ-55375515 Dose Level 2; Drug: JNJ-55375515 Dose Level 4; Drug: JNJ-55375515 Dose Level 6; Drug: Placebo
- Part 2: JNJ-55375515 and placebo (Experimental): Participants will randomly be assigned to one of four treatment sequences 1, 2, 3 or 4. In the first 3 sequences, participants will receive 2 doses of JNJ-55375515 and placebo. Participants assigned to sequence 4 will receive placebo only in all periods. 3 dose levels will be tested in Part 2 based on Part 1 and will not exceed those evaluated in Part 1. A wash-out period of at least 10 days will be maintained between study drug administrations in period 1, 2, 3 and 4. In period 4 (open-label pharmacokinetic (PK) assessment period) participants will be randomly assigned to one of two dose levels tested in periods 1 to 3.
  Interventions: Drug: Placebo; Drug: JNJ-55375515

INTERVENTIONS:
Drug: JNJ-55375515 Dose Level 1 — Participants will receive JNJ-55375515 orally at a Dose level 1 in Part 1 of study.
  Arms: Part 1 (Panel 1): JNJ-55375515 and placebo
Drug: JNJ-55375515 Dose Level 2 — Participants will receive JNJ-55375515 orally at a Dose level 2 in Part 1 of study.
  Arms: Part 1 (Panel 2): JNJ-55375515 and placebo
Drug: JNJ-55375515 Dose Level 3 — Participants will receive JNJ-55375515 orally at a Dose level 3 in Part 1 of study.
  Arms: Part 1 (Panel 1): JNJ-55375515 and placebo
Drug: JNJ-55375515 Dose Level 4 — Participants will receive JNJ-55375515 orally at a Dose level 4 in Part 1 of study.
  Arms: Part 1 (Panel 2): JNJ-55375515 and placebo
Drug: JNJ-55375515 Dose Level 5 — Participants will receive JNJ-55375515 orally at a Dose level 5 in Part 1 of study.
  Arms: Part 1 (Panel 1): JNJ-55375515 and placebo
Drug: JNJ-55375515 Dose Level 6 — Participants will receive JNJ-55375515 orally at a Dose level 6 in Part 1 of study.
  Arms: Part 1 (Panel 2): JNJ-55375515 and placebo
Drug: Placebo — All participants will receive matching placebo orally in Part 1 and Part 2 of the study.
Drug: JNJ-55375515 — Participants will receive JNJ-55375515 as per the assigned treatment in Part 2.
  Arms: Part 2: JNJ-55375515 and placebo

SUMMARY:
The purpose of this study is to assess safety and tolerability of day-time and night-time dosing of JNJ-55375515 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 and 30 kilogram / square meter (kg/m^2) inclusive (BMI=weight/height^2)
* Participant must be healthy based on clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, coagulation or urinalysis are outside the normal reference ranges, retesting of an abnormal lab value (s) that may lead to exclusion will be allowed once during the screening phase. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the investigator, are acceptable
* Participant must be healthy based on physical and neurological examination, medical history, vital signs, and 12-lead Electrocardiography (ECG) [including QTcF less than or equal to (<=) 450 millisecond (msec)] performed at screening, admission to the clinical unit and pre dose on Day 1 of Period 1. Abnormalities, which are not considered to be of clinical significance by the investigator, are acceptable. The presence of Left Bundle Branch Block (LBBB), AV Block (second degree or higher), or a permanent pacemaker or implantable cardioverter defibrillator [ICD] will lead to exclusion
* Non-smoker (not smoked for 3 months prior to screening)
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study drug, in addition to the highly effective method of contraception, a man who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (for example, condom with spermicidal foam/gel/film/cream/suppository); who is sexually active with a woman who is pregnant must use a condom; must agree not to donate sperm

Exclusion Criteria:

* History of or current significant medical illness including (but not limited to psychotic, bipolar, major depressive, or anxiety disorder)
* Cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the participant
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies
* Participant has a history of or current vestibular disease including (but not limited to) Meniere's disease, benign paroxysmal positional vertigo (BPPV), vestibular neuronitis, vestibular schwannoma or vestibular migraine
* Only for part 2: Has a current diagnosis or history of narcolepsy, central sleep apnea, sleep related hypoventilation, circadian rhythm sleep-wake disorders, substance/medication induced sleep disorder or parasomnias (non-rapid eye movement sleep arousal disorders, nightmare disorder, rapid eye movement sleep behavior disorder); obstructive sleep apnea/hypopnea (apnea/hypopnea index greater than (>)10) or restless legs syndrome (periodic leg movements with arousal index >15); night-shift worker or significantly shifted diurnal activity pattern (it is expected that eligible participant normally wake up between 6:00 am - 8:00 am and go to bed between 10:00 pm - 12:00 am); usual bedtime outside of 10:00 pm and 12:00 am and taking, on average, less than 6 hours or more than 9 hours of bed rest

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Part 1 (Day-Time Dosing): Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Week 8
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Part 2 (Night-Time Dosing): Number of Participants with AEs as a Measure of Safety and Tolerability | Up to Week 9
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.

SECONDARY OUTCOMES:
Slow Wave Activity Recorded by the Electroencephalogram (EEG) | Pre-dose, 1 hour (h), 2h, and 4h post dose on Day 1
  The Effect of JNJ-55375515 on slow wave activity recorded by the electroencephalogram (EEG) will be evaluated. EEG recordings are made using gold electrodes, fixed at Midline Frontal Electrode (Fz), Midline Central Electrode (Cz), Midline Parietal Electrode (Pz) and Midline Occipital Electrode (Oz), with the same common ground electrode as for the eye movement registration (international 10/20 system). Per session eight consecutive blocks of eight seconds are recorded. For each lead, fast Fourier transform analysis will be performed to obtain the sum of amplitudes in the very low (0.5-2 Hertz [Hz]), delta- (2-4 Hz), theta (4-7.5 Hz), alpha- (7.5-13.5 Hz), beta- (13.5-35 Hz), and gamma-(35-48.9 Hz) frequency ranges. The total test will last approximately 2 minutes.
Part 1: PD of JNJ-55375515 as Assessed by Heart Rate Variability (HRV) | Pre-dose (Day 1) up to 24 hours post dose
  Heart rate variability (HRV) is the physiological phenomenon of variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval. HRV will be derived from Holter recordings. Holter recordings will start pre dose on Day 1 of each period in Part 1 and continue for 24 hours. Measurements will be made at rest (during 5 minutes) and HRV parameters will be derived from these 5-minute recordings and from the 24-hour recordings.
Part 1: Saccadic Reaction Time (RT) as Measured by Saccadic Eye Movements | Pre-dose, 1 h, 2h, and 4h post dose on Day 1
  Saccadic eye movements will be recorded to measure saccadic reaction time (RT). The recording and analysis of saccadic eye movements is performed using a computer-based system for sampling and analysis of eye movements. In a typical test system, electrodes are applied on the forehead and beside the lateral canthi of both eyes of the participant for registration of the electro-oculographic signals. Head movements are restrained using a fixed head support. The target consists of a moving dot that is displayed on a computer screen. Fifteen saccades are recorded with inter-stimulus intervals varying randomly between 3 and 6 seconds. Average values of latency (reaction time) of all correct saccades will be assessed.
Part 1: Saccadic Peak Velocity (SPV) as Measured by Saccadic Eye Movements | Pre-dose, 1h, 2h, and 4h post dose on Day 1
  Saccadic eye movements will be recorded to measure saccadic peak velocity (SPV). The recording and analysis of saccadic eye movements is performed using a computer-based system for sampling and analysis of eye movements. In a typical test system, electrodes are applied on the forehead and beside the lateral canthi of both eyes of the participant for registration of the electro-oculographic signals. Head movements are restrained using a fixed head support. The target consists of a moving dot that is displayed on a computer screen. Fifteen saccades are recorded with inter-stimulus intervals varying randomly between 3 and 6 seconds. Average values of saccadic peak velocity of all correct saccades will be assessed.
Part 1: Change from Baseline in Body Sway | Baseline, 1h, 2h, and 4h post dose on Day 1
  The body sway meter allows measurement of body movements in a single plane, providing a measure of postural stability. Body sway may be measured with a pot string meter (Celesco) based on the Wright ataxiameter or platform. Participants will be instructed to wear a pair of comfortable, low-heeled shoes on each session. The total period of body-sway measurement will be 2 minutes.
Part 1 and 2: PD as Assessed by Karolinska Sleepiness Scale (KSS) Score | Part 1: Pre-dose, 1h, 3h, and 8h post dose on Day 1; Part 2: Pre-dose (Day 1) and 8h post dose (Day 2)
  The KSS is a patient reported assessment of drowsiness level at the time of scale administration. This scale is focused mainly on the propensity to fall asleep and has a high validity in assessing sleepiness. It consists of a 9-point Likert scale with response options from: 1=very alert, 3=alert, 5=neither alert nor sleepy, 7=sleepy (but not fighting sleep), 9=very sleepy (fighting sleep).
Part 1: Change from Baseline in Bond and Lader Visual Analogue Scale (B&L VAS) Score | Baseline, 1h, 2h, and 4h post dose on Day 1
  The Bond and Lader Visual Analogue Scale consists of sixteen 100 millimeter (mm) visual analog scales anchored by antonyms (example, Alert-Drowsy, Lethargic-Energetic, etc). Scores will be combined to form three mood factors: alertness, calmness, and contentedness.
Part 1 and 2: Change from Baseline in Cortisol Levels | Part 1: Baseline, 0.5h, 1h, 2h, 3h, 4h, 5h 45minutes (m), 6h, 6h 05m, 6h 25m, 6h 30m, 6h 50m, 6h 55m, 7h 15m, 7h 35m, 8h, 12h and 24h post dose on Day 1; Part 2: Baseline, 0.5h, 1h, 2h (Day 1 or 2), 3h, 4h, 6h, 8h, 12h and 24h post dose on Day 2
  To establish diurnal levels of cortisol levels, repeated serum samples will be obtained throughout the Day 1 of each period. The diurnal cortisol levels will be explored to further clarify the effect of the compound on the hypothalamic-pituitary-adrenal-axis.
Part 1: PD as Assessed by Probabilistic Instrumental Learning Task (PILT) | Pre-dose, 3h, and 8h post dose on Day 1
  In this motivational processing task, participants with depressive symptoms may show a lower response bias towards a reward compared to healthy participants. The PILT allows the objective assessment of participants propensity to modulate behavior as a function of reward.
Part 1: PD as Assessed by Cognitive Test Battery: International Shopping List Test | Pre-dose, 3h, and 8h post dose on Day 1
  The International Shopping List Test is a measure of Verbal Memory-Learning. The test measures total number of correct responses remembering the 16-word list on three consecutive learning trials. Higher score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: Groton Maze Learning Task | Pre-dose, 3h, and 8h post dose on Day 1
  Groton Maze Learning Task is a measure of Executive Function and Spatial Learning. The test measures total number of errors made while locating and learning 28 step pathway hidden beneath a 10*10 grid on 5 consecutive trials during a single session. Lower score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: Social Emotional Cognition Task | Pre-dose, 3h, and 8h post dose on Day 1
  To evaluate social and emotional cognition, a series of tests will be used to quantify both the ability to empathize and understand the emotions of others, and the ability to interpret their thoughts and intentions. A classical test involves the presentation of facial expressions and is asked to choose which word best describes what the person in the image is thinking or trying.
Part 1: PD as Assessed by Cognitive Test Battery: Detection Task | Pre-dose, 3h, and 8h post dose on Day 1
  Detection task is a measure of Psychomotor Function. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: Identification Task | Pre-dose, 3h, and 8h post dose on Day 1
  Identification task is a measure of Attention. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: one Back Task | Pre-dose, 3h, and 8h post dose on Day 1
  One back task is a measure of Working Memory. The test measures speed of performance; mean of the log10 transformed reaction times for correct responses. Lower score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: International Shopping List Test - Delayed Recall | Pre-dose, 3h, and 8h post dose on Day 1
  International shopping list test - Delayed Recall is a measure of Delayed Verbal Memory. The test measures total number of correct responses recalling the 16 words learned previously after a delay. Higher score indicates better performance.
Part 1: PD as Assessed by Cognitive Test Battery: Groton Maze Learning - Delayed Recall | Pre-dose, 3h, and 8h post dose on Day 1
  Groton Maze Learning - Delayed recall is a measure of Delayed Spatial Memory. The test measures number of errors made while locating 28 step pathway hidden beneath a 10*10 grid after a delay. Lower score indicates better performance.
Part 1: Evoked Stress Response as Assessed by Induced Stress | 6h 30m to 6h 50m post dose on Day 1
  The induced stress test consists of a highly demanding computer task that is performed for 20 minutes.
Part 2: Latency to Persistent Sleep (LPS) by 8-hour Overnight Polysomnography | 0 hour (Day 1) up to 8 Hour (Day 2)
  LPS is the time in minutes from 'lights out' that marks the starting of total recording time to the first epoch scored as sleep.
Part 2: Total Time Spent in Deep Sleep (Duration of Slow Wave Sleep) - Stage 3 Sleep by 8-Hour Overnight Polysomnography | 0 hour (Day 1) up to 8 Hour (Day 2)
  Polysomnographic recordings will be used to determine the total time spent in deep sleep (duration of slow wave sleep) -stage 3 sleep by 8-hour overnight.
Part 2: Time in bed by 8-hour Overnight Polysomnography | 0 hour (Day 1) up to 8 Hour (Day 2)
  Polysomnographic recordings will be used to determine the time in bed by 8-hour overnight.
Part 2: Cognitive Test Battery: Continuous Paired Associate Learning Task (CPAL) | -7 hour (Day 1), 17 hour (Day 2)
  The Continuous Paired Associate Learning (CPAL) test will be used to assess whether JNJ-55375515 will improve performance of complex cognitive tasks. CPAL assess Visual episodic memory (associate learning) cognitive domain. In this task, participants must learn a series of associations between a set of difficult to verbalize patterns (amoeba) and locations. In healthy adults, 14 pattern/location associations must be learned. In the presentation phase of the task the pattern appears at the location and the participant is required to acknowledge that they have seen the pattern by touching the location at which it appears. Patterns are presented in random order. In the learning phase of the task, participants must place each of the 14 patterns in their correct locations. They must do this in 10 rounds. Number of errors made in correctly placing each of the four patterns in their location four times. (Lower score = better performance).
Part 1 and 2: Maximum Observed Plasma Concentration (Cmax) | Part 1: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, and 96h post dose; Part 2: Pre dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 46h, 70h, and 94h post dose
  Cmax is the maximum observed plasma concentration.
Part 1 and 2: Time to Reach Maximum Observed Plasma Concentration (Tmax) | Part 1: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, and 96h post dose; Part 2: Pre dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 46h, 70h, and 94h post dose
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Part 1 and 2: Area Under the Plasma Concentration-Time Curve from Time 0 to Time of the Last Quantifiable Concentrations (AUC[0-last]) | Part 1: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h, 72h, and 96h post dose; Part 2: Pre-dose, 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 46h, 70h, and 94h post dose
  AUC(0-last) is area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands